CLINICAL TRIAL: NCT04787029
Title: Effect of Prophylactic Medical Compression Therapy on the Reduction of Breast Cancer-related Lymphedema in Patients With Adjuvant Docetaxel Chemotherapy: a Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMC 2020-11-051
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prophylactic medical compression therapy group (Experimental): This study provides medical compression stockings from the start date of Docetaxel administration for patients who have undergone mastectomy and axillary lymphectomy for breast cancer, and who are planning to receive Docetaxel adjuvant chemotherapy. The intervention group wears medical compression stockings for upper limbs with a pressure level of 1 (15-21mmHg) during the day from the start of docetaxel administration to 3 months after the end of administration.
  Basic education of upper limb exercises (joint motion range enhancement exercises and upper limb muscle pumping exercises) is provided to both the intervention group and the control group.
  Interventions: Device: Medical compression stocking (medical device name: mediven Harmony 734 (compression class1 AG armsleeve or with wide(735))
- control group (No Intervention): The control group proceeds as an observation, but interventions such as providing stockings in the event of lymphedema are performed.
  Basic education of upper limb exercises (joint motion range enhancement exercises and upper limb muscle pumping exercises) is provided to both the intervention group and the control group.

INTERVENTIONS:
Device: Medical compression stocking (medical device name: mediven Harmony 734 (compression class1 AG armsleeve or with wide(735)) — Compression stockings worn on the arm or partial swelling of the hand after trauma or surgery.
  Arms: prophylactic medical compression therapy group

SUMMARY:
In this study, the purpose of this study is to investigate whether prophylactic medical compression therapy in breast cancer patients receiving docetaxel adjuvant chemotherapy could reduce the incidence and severity of lymphedema in the upper limbs that received axillary lymph node resection (sentinel lymph node biopsy or axillary lymph node dissection).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent radical mastectomy and sentinel lymphctomy or axillary lymphectomy after diagnosis of unilateral breast cancer
2. Patients who are scheduled for adjuvant chemotherapy including Docetaxel after surgery
3. Patients aged 19 to 70
4. Patients who can understand the contents of this study and obtain consent

Exclusion Criteria:

1. Patients with a history of breast-related surgery prior to this breast cancer surgery
2. Patients with metastases to other organs
3. Patients who have undergone neoadjuvant chemotherapy or have previously received radiation therapy
4. Patients with systemic diseases that may not be able to conduct clinical research
5. Patients with skin diseases who cannot receive medical compression treatment

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence rate of lymphedema (%) | The cumulative incidence of lymphedema during the entire primary observation period
  The cumulative incidence rate of lymphedema The cumulative incidence of lymphedema during the entire primary observation period (Enrollment (pre-docetaxcel), mid-docetaxcel(up to 20 weeks), Post-docetaxcel 1month, Post-docetaxcel 3month, Post-docetaxcel, 6month, Post-docetaxcel, 1year, Post-docetaxcel, 1.5year, Post-docetaxcel 2year) permanent lymphedema criteria:
  1. excess limb volume (≥10%, forearm or whole arm)
  2. excess limb volume (<10%, forearm or whole arm, If there is regional lymphedema suitable for lymphatic territory and a Lymphedema specialist makes a clinical diagnosis)
Severity of lymphedema - percentage of excess limb volume (PCEV, ml) | Time of occurrence of lymphedema during the follow-up period
  Limb lymphedema volumes were measured using the electronic volumeter device (Perometer; Pero-System, Wuppertal, Germany), which is an optoelectronic instrument for measuring limb volume and circumferences.
  PCEV (%) = [(volume of affected limb - volume of unaffected limb) / volume of unaffected limb] × 100 Volume comparison between groups at the onset of lymphedema during the follow-up period (Enrollment (pre-docetaxcel), mid-docetaxcel(up to 20 weeks), Post-docetaxcel 1month, Post-docetaxcel 3month, Post-docetaxcel, 6month, Post-docetaxcel, 1year, Post-docetaxcel, 1.5year, Post-docetaxcel 2year)

SECONDARY OUTCOMES:
ECW/TBW ratio (%) of whole body (body water analysis result) | Enrollment (pre-docetaxcel), mid-docetaxcel(up to 20 weeks), Post-docetaxcel 1month, Post-docetaxcel 3month, Post-docetaxcel, 6month, Post-docetaxcel, 1year, Post-docetaxcel, 1.5year, Post-docetaxcel 2year
  This ratio will be measured using Inbody scale (S10) on each observation period and this trend will be analyzed by time, group and interaction

CONTACTS AND LOCATIONS:
Overall Officials: JIHYE HWANG, Professor, Study Chair — Physical & Rehabilitation Medicine Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided